CLINICAL TRIAL: NCT02648373
Title: Effect of a Patient Education Intervention for Patients With Low Back Pain Referred to Physical Therapy
Brief Title: Patient Education for Patients With Back Pain Referred to Physical Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Julie Fritz, Ph.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00072901
Record Dates: First submitted 2015-05-27; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental): Patients receive an educational video about low back pain based on the Consumer Reports Choosing Wisely recommendation for patients with back pain to avoid early imaging and remain as active as possible. After the video the evaluator and patient discussed key themes from the video and the patient was able to ask any questions. Previously scheduled physical therapy then began with treatment at the therapist's discretion.
  Interventions: Behavioral: Patient Education
- Control (Active Comparator): Previously scheduled physical therapy was provided with treatment at the therapist's discretion. No educational intervention was provided before beginning physical therapy
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Patient Education — An educational video was watched based on Consumer Reports Choosing Wisely patient education supporting the recommendation that imaging is not helpful early for low back pain and the best strategy is to remain as active as possible. Key themes were discussed with a physical therapist and the patient's questions were answered.
  Arms: Education
Other: Control — Patients receive no additional intervention. They will begin physical therapy and receive care at the therapist's discretion.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate patients with low back pain who are scheduled to begin physical therapy but have not yet had their first appointment to better understand their beliefs and attitudes and to evaluate the effects of an educational session about low back pain.

DETAILED DESCRIPTION:
The investigators will conduct a randomized trial to examine the effectiveness of a patient education session provided prior to beginning physical therapy on outcomes of usual physical therapy for acute/sub-acute low back pain patients. The study compares two groups, one group will be treated with usual physical therapy with no pre-treatment education and the other group will also receive the pre-treatment. Patients will be followed after 6 weeks and 3 months. Physical therapy care is left to the discretion of the physical therapist in conjunction with the patient. Outcomes will include pain and disability, and patients attitude and believes (pain catastrophizing, fear avoidance behavior). The overall hypothesis is that the additional educational treatment may address and improve pain, disability and fear.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of non-specific low back pain scheduled to receive outpatient physical therapy
* age 18-60
* duration of current symptoms < 8weeks
* referred to physical therapy from a non-surgeon provider
* no treatment received for low back pain in past year other than physician office visits.

Exclusion Criteria:

* Diagnosis provided by the referral source indicating a specific pathoanatomical source for LBP including fracture, spondylolesthesis, ankylosing spondylitis, radiculopathy
* any red flags in the patient's general medical screening questionnaire (i.e. tumor, metabolic diseases etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 6 weeks
  Self-report measure of low back pain-related disability
Pain as measured by the Numeric Pain Rating Scale | 6 weeks
  Self-report measure of pain intensity on 0-10 rating scale

SECONDARY OUTCOMES:
Fear Avoidance beliefs Questionnaire | baseline, 6 weeks, 3 months
  Self-report measure of fear avoidance beliefs about physical activity and work
Pain Catastrophizing Scale | baseline, 6 weeks, 3 months
  Self-report measure of pain catastrophizing beliefs
Pain Beliefs Questionnaire | baseline, 6 weeks, 3 months
  Self-report questionnaire used to measure patients' beliefs about the causes and consequences of pain with 2 subscales: organic (i.e, biomedical) and psychological.
Global Rating of Change | 6 weeks, 3 months
  Self-report global rating of improvement in condition since baseline assessed on 0-15 scale
Physical Therapy Visits: Number of physical therapy episodes attended after baseline | 6 weeks, 3 months
  Number of physical therapy episodes attended after baseline
Treatment Self-Regulation Questionnaire | baseline, 6 weeks, 3 months
  Self-report questionnaire examining motivations to attend physical therapy
Hospital Anxiety and Depression Scale | baseline, 6 weeks, 3 months
  Self-report questionnaire assessing anxiety and depression in separate sub-scales
Oswestry Disability Scale | baseline, 3 months
  Self-report measure of low back pain-related disability
Numeric Pain Rating | baseline, 3 months
  Self-report measure of pain intensity on 0-10 scale

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Utah Healthcare System, Salt Lake City, Utah, United States